CLINICAL TRIAL: NCT01205061
Title: A Pivotal USA Randomized, Evaluator-blinded, Active-controlled, Multi-center, Split-face Comparison Study of Emervel® Deep Lidocaine Versus Juvederm® Ultra Plus in the Treatment of Moderate to Severe Facial Wrinkles and Folds
Brief Title: Emervel® Deep Lidocaine vs. Juvederm® Ultra Plus in Treatment of Moderate to Severe Facial Wrinkles and Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.06.CIP.18159
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-07

CONDITIONS: Skin Wrinkling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Emervel Deep Lidocaine (Experimental): NLFs (Nasolabial Folds) were injected with Emervel Deep Lidocaine (20 mg/mL with 0.3% lidocaine).
  Interventions: Device: Emervel Deep Lidocaine
- Juvederm Ultra Plus (Active Comparator): NLFs were injected with Juvéderm Ultra Plus (24 mg/mL).
  Interventions: Device: Juvederm Ultra Plus

INTERVENTIONS:
Device: Emervel Deep Lidocaine — 20 mg/mL + 0.3% lidocaine
  Arms: Emervel Deep Lidocaine
Device: Juvederm Ultra Plus — 24mg/mL
  Arms: Juvederm Ultra Plus

SUMMARY:
The purpose of the study was to compare the effectiveness and safety of Emervel Deep Lidocaine versus Juvederm Ultra Plus in the treatment of moderate to severe facial wrinkles and folds.

DETAILED DESCRIPTION:
This was a randomized, evaluator-blinded, active-controlled, multi-center, split-face comparison study of Emervel Deep Lidocaine versus Juvederm Ultra Plus in the treatment of moderate to severe facial wrinkles and folds. Two physicians, an Unblinded Injecting Investigator and a Blinded Evaluating Investigator, were required at each study center. The Unblinded Injecting Investigator was different from the Blinded Evaluating Investigator.

ELIGIBILITY:
Inclusion Criteria:

* The subject was a male or female 18 years of age or older
* The subject had bilateral nasolabial folds that, in the opinion of both the blinded evaluating investigator and the unblinded injecting investigator, was corrected with an injectable dermal implant
* The subject had the same Wrinkle Severity Rating Scale (WSRS) score of 3 or 4 (moderate or severe) for each nasolabial fold

Exclusion Criteria:

* The subject had active skin disease or inflammation on or near a nasolabial fold that, in the principal investigator's opinion, would interfere with the study device injections and/or study assessments.
* The subject had a history of sensitivity to hyaluronic acid
* The subject had a history of sensitivity to lidocaine or other amide type anesthetics
* The subject was, in the principal investigator's opinion, at undue risk based on the precautions, warnings and contraindications for local lidocaine anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2010-09-27 (Actual); Primary Completion 2011-06-20 (Actual); Study Completion 2012-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, M.D., Study Chair — Galderma R&D
Locations (11):
- United States (11):
  - Galderma research site, Los Angeles, California
  - Galderma research site, San Francisco, California
  - Galderma research site, New Haven, Connecticut
  - Galderma research site, Miami Beach, Florida
  - Galderma research site, Snellville, Georgia
  - Galderma research site, Hunt Valley, Maryland
  - Galderma research site, Warren, Michigan
  - Galderma research site, White Plains, New York
  - Galderma research site, Charlotte, North Carolina
  - Galderma research site, Nashville, Tennessee
  - Galderma research site, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 11 sites in the United States from 27 September 2010 to 12 January 2012.
Pre-assignment Details: A total of 184 participants were screened, of which 162 participants received treatment in this study.
Groups:
- All Participants: Participants were randomized to receive either Emervel Deep Lidocaine (20 milligram per milliliter [mg/mL] with 0.3% lidocaine) injection in the left nasolabial fold (NLF) and Juvederm Ultra Plus (24 mg/mL) injection in to the right NLF or Juvederm Ultra Plus (24 mg/mL) injection in the left NLF and Emervel Deep Lidocaine (20 mg/mL with 0.3% lidocaine) injection in the right NLF.
Period: Overall Study
Arm/Group | All Participants
Started | 162
Emervel Deep Lidocaine in Left NLF Followed by Juvederm Ultra in Right NLF | 80
Juvederm Ultra in Left NLF Followed by Emervel Deep Lidocaine in Right NLF | 82
Completed | 136
Not Completed | 26
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 11
Not completed — Clinical Investigational Plan Violation | 1
Not completed — Lost to Follow-up | 9
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat population included all participants who were randomized and received an injection on both treatment sides.
Groups:
- Emervel Deep Lidocaine in Left NLF Followed by Juvederm Ultra Plus in Right NLF: Participants received Emervel Deep Lidocaine (20 mg/mL with 0.3% lidocaine) injection into the left NLF and Juvéderm Ultra Plus (24 mg/mL) in the right NLF.
- Juvederm Ultra Plus in Left NLF Followed by Emervel Deep Lidocaine in Right NLF: Participants received Juvéderm Ultra Plus (24 mg/mL) injection into the left NLF and Emervel Deep Lidocaine (20 mg/mL with 0.3% lidocaine) injection in the right NLF.
- Total: Total of all reporting groups
Arm/Group | Emervel Deep Lidocaine in Left NLF Followed by Juvederm Ultra Plus in Right NLF | Juvederm Ultra Plus in Left NLF Followed by Emervel Deep Lidocaine in Right NLF | Total
Number analyzed (Participants) | 80 | 82 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (9.29) | 54.0 (8.09) | 53.7 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 78 | 156
  Male | 2 | 4 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 63 | 66 | 129
  Race: Black | 9 | 11 | 20
  Race: Hispanic | 5 | 5 | 10
  Race: Other | 3 | 0 | 3
Skin Type [Count of Participants; unit: Participants] — Skin Type I = White; very fair, red or blonde hair blue eyes; freckles; Always burns, never tans Skin Type II = White, fair, red or blond hair; blue, hazel or green eyes; Usually burns, tans with difficulty Skin Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans Skin Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease Skin Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily Skin Type VI = Black; Never burns, tans very easily
  Participants
    Type I | 1 | 5 | 6
    Type II | 16 | 12 | 28
    Type III | 30 | 37 | 67
    Type IV | 18 | 16 | 34
    Type V | 11 | 8 | 19
    Type VI | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Wrinkle Severity Rating Scale (WSRS) at Week 24 After Final Initial Injection
Description: WSRS is a validated 5-point reference scale with photographs that classifies deep facial wrinkles (nasolabial folds). WSRS represents clinically meaningful change in NLF severity from the adjacent grades where 1= absent (no visible fold; continuous skin line), 2 = mild (shallow but visible fold with a slight indentation; minor facial feature; implant expected to produce a slight improvement in appearance), 3 = excellent (correction is expected from injectable implant), 4 = severe (very long and deep folds; prominent facial feature; less than 2 mm visible fold when stretched; significant improvement expected from injectable implant), 5 = extreme (extremely deep and long folds, detrimental to facial appearance; 2 to 4 millimeter (mm) visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 24 after final initial injection (Week 24 for participants without touch-up injection, Week 27 for participants with touch-up injection at Week 3)
Population: Intent to Treat (ITT) population included participants who were randomized and received an injection on both treatment sides.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Emervel Deep Lidocaine: NLFs were injected with Emervel Deep Lidocaine (20 mg/mL with 0.3% lidocaine).
Arm/Group | Emervel Deep Lidocaine | Juvederm Ultra Plus
Number analyzed (Participants) | 162 | 162
Score on a scale | -1.1 (0.75) | -1.1 (0.68)

2. Secondary Outcome: Mean Change From Baseline in Wrinkle Severity Rating Score (WSRS) at Week 3 After Final Initial Injection
Description: WSRS is a validated 5-point reference scale with photographs that classifies deep facial wrinkles (nasolabial folds). WSRS represents a clinically meaningful change in nasolabial fold severity from the adjacent grades where 1 = absent (no visible fold; continuous skin line), 2 = mild (shallow but visible fold with a slight indentation; minor facial feature; implant is expected to produce a slight improvement in appearance), 3 = excellent (correction is expected from injectable implant), 4 = severe (very long and deep folds; prominent facial feature; less than 2 mm visible fold when stretched; significant improvement is expected from injectable implant), 5 = extreme (extremely deep and long folds, detrimental to facial appearance; 2 to 4 mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 3 after final initial injection (Week 3 for participants without touch-up injection, Week 6 for participants with touch-up injection at Week 3)
Population: ITT population included participants who were randomized and received an injection on both treatment sides.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Emervel Deep Lidocaine | Juvederm Ultra Plus
Number analyzed (Participants) | 162 | 162
Score on a scale | -1.6 (0.62) | -1.6 (0.64)

3. Secondary Outcome: Mean Change From Baseline in Wrinkle Severity Rating Score (WSRS) at Week 12 After Final Initial Injection
Description: as for outcome 2
Time Frame: Baseline, Week 12 after final initial injection (Week 12 for participants without touch-up injection, Week 15 for participants with touch-up injection at Week 3)
Population: ITT population included participants who were randomized and received an injection on both treatment sides.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Emervel Deep Lidocaine | Juvederm Ultra Plus
Number analyzed (Participants) | 162 | 162
Score on a scale | -1.3 (0.70) | -1.3 (0.74)

4. Secondary Outcome: Mean Change From Baseline in Wrinkle Severity Rating Score (WSRS) at Week 36 After Final Initial Injection
Description: as for outcome 2
Time Frame: Baseline, Week 36 after final initial injection (Week 36 for participants without touch-up injection, Week 39 for participants with touch-up injection at Week 3)
Population: ITT population included participants who were randomized and received an injection on both treatment sides.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Emervel Deep Lidocaine | Juvederm Ultra Plus
Number analyzed (Participants) | 162 | 162
Score on a scale | -1.1 (0.67) | -1.1 (0.68)

5. Secondary Outcome: Mean Change From Baseline in Wrinkle Severity Rating Score (WSRS) at Week 48 After Final Initial Injection
Description: WSRS is a nasolabial fold severity from the adjacent grades where 1 = absent (no visible fold; continuous skin line), 2 = mild (shallow but visible fold with a slight indentation; minor facial feature; implant is expected to produce a slight improvement in appearance), 3 = excellent (correction is expected from injectable implant), 4 = severe (very long and deep folds; prominent facial feature; less than 2 mm visible fold when stretched; significant improvement is expected from injectable implant), 5 = extreme (extremely deep and long folds, detrimental to facial appearance; 2 to 4 mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 48 after final initial injection (Week 48 for participants without touch-up injection, Week 51 for participants with touch-up injection at Week 3)
Population: ITT population included participants who were randomized and received an injection on both treatment sides.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Emervel Deep Lidocaine | Juvederm Ultra Plus
Number analyzed (Participants) | 162 | 162
Score on a scale | -0.8 (0.66) | -0.9 (0.66)

6. Secondary Outcome: Mean Change From Baseline in Participant Self-Assessment of Wrinkle Severity at Week 24 After Final Initial Injection
Description: Participants self-assessment was measured by using a wrinkle severity scale with 1 being absent and 5 being extreme. Each participant was to perform an assessment of the wrinkle severity based on self-assessment score: 1= Absent (No visible fold; continuous skin line), 2= Mild (Shallow but visible fold with a slight indentation), 3= Moderate (Moderately deep folds), 4= Severe (Very long and deep fold), 5= Extreme (Extremely deep and long folds). A negative change from baseline indicates improvement.
Time Frame: as for outcome 1
Population: ITT population included participants who were randomized and received an injection on both treatment sides.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Emervel Deep Lidocaine | Juvederm Ultra Plus
Number analyzed (Participants) | 162 | 162
Score on a scale | -1.2 (0.91) | -1.3 (0.75)

7. Secondary Outcome: Participant Pain Assessment After the Initial Injection
Description: Participant pain severity for each NLF was assessed at time 0, 15, 30, 45, 60 minutes and 24 hours after the initial injection using an 11-point Numeric Pain Intensity Scale (NPIS).The NPIS was a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with 0 is no pain and 10 is the worst possible pain where a lower score correlates to better outcome for pain.
Time Frame: At 0 ,15, 30, 45, 60 minutes and 24 hours after the initial injection (Baseline)
Population: ITT population included participants who were randomized and received an injection on both treatment sides. Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given timepoints.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Emervel Deep Lidocaine | Juvederm Ultra Plus
Number analyzed (Participants) | 162 | 162
Score on a scale
  At 0 Minutes | 3.1 (2.1) | 5.3 (2.3)
  At 15 Minutes | 0.5 (0.9) | 1.8 (1.8)
  At 30 Minutes | 0.2 (0.6) | 1.0 (1.5)
  At 45 Minutes | 0.1 (0.4) | 0.5 (1.0)
  At 60 Minutes | 0.1 (0.3) | 0.3 (0.8)
  At 24 Hours: number analyzed (Participants) | 160 | 160
  At 24 Hours | 0.9 (1.5) | 0.9 (1.6)

8. Secondary Outcome: Participant Pain Assessment After the Initial Touch-up Injection
Description: Participant pain severity for each NLF was assessed at time 0, 15, 30, 45, 60 minutes and 24 hours after the initial injection using NPIS. The NPIS was a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with 0 is no pain and 10 is the worst possible pain where a lower score correlates to better outcome for pain.
Time Frame: At 0, 15, 30, 45, 60 minutes and 24 hours after the Initial Touch-up Injection (At 3 weeks after initial injection)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Emervel Deep Lidocaine | Juvederm Ultra Plus
Number analyzed (Participants) | 86 | 80
Score on a scale
  At 0 Minutes | 3.3 (2.2) | 4.8 (2.4)
  At 15 Minutes | 0.7 (1.2) | 1.2 (1.6)
  At 30 Minutes | 0.3 (0.7) | 0.5 (1.0)
  At 45 Minutes | 0.1 (0.4) | 0.2 (0.7)
  At 60 Minutes | 0.1 (0.3) | 0.1 (0.5)
  At 24 Hours: number analyzed (Participants) | 84 | 79
  At 24 Hours | 0.5 (0.9) | 0.6 (1.3)

9. Secondary Outcome: Number of Participants With Adverse Event (AEs)
Description: AE was defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with the study drug. Number of participants with AEs were reported. Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."
Time Frame: From start of study drug administration up to 62 weeks
Population: Safety population included all participants who received at least one injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Emervel Deep Lidocaine | Juvederm Ultra Plus
Number analyzed (Participants) | 162 | 162
Participants | 66 | 67

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 62 weeks
Description: The safety population included all participants who received at least one injection.
Arm/Group | Emervel Deep Lidocaine | Juvederm Ultra Plus
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/162
Serious Adverse Events (participants affected / at risk) | 7/162 | 7/162
Other Adverse Events (participants affected / at risk) | 16/162 | 16/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Emervel Deep Lidocaine (N=162) | Juvederm Ultra Plus (N=162)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 — Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 — Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 — Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."
Herpes Zoster (Infections and infestations) | 1 | 1 — Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."
Diarrhoea infections (Infections and infestations) | 1 | 1 — Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 — Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."
Lumbar Spinal stenosis (Infections and infestations) | 1 | 1 — Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 1 — Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Emervel Deep Lidocaine (N=162) | Juvederm Ultra Plus (N=162)
Upper respiratory tract infection (Infections and infestations) | 6 | 6
Sinusitis (Infections and infestations) | 5 | 5
Migraine (Nervous system disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other